CLINICAL TRIAL: NCT02508935
Title: A Phase 4, Open-Label Study of the Pharmacokinetics and Safety of XARTEMIS® XR (7.5 Oxycodone Hydrochloride/325 mg Acetaminophen) in Postsurgical Adolescent Subjects (Ages 12 to 17) With Moderate to Severe Acute Pain
Brief Title: Pharmacokinetics (PK) and Safety Study of XARTEMIS® XR in Postsurgical Adolescent Subjects With Moderate to Severe Acute Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Business decision
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNK15000300
Record Dates: First submitted 2015-06-17; First posted 2015-07-27 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2018-05

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — oxycodone-acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- XARTEMIS XR (Experimental): All participants received XARTEMIS XR
  Interventions: Drug: XARTEMIS XR

INTERVENTIONS:
Drug: XARTEMIS XR — XARTEMIS XR [7.5 mg oxycodone hydrochloride and 325 mg acetaminophen (APAP)] Extended-Release Tablets

SUMMARY:
Phase 4, multicenter, open-label, multiple-dose study of the pharmacokinetics (PK) and safety of XARTEMIS XR in postsurgical adolescent subjects aged 12 to 17 years with moderate to severe acute pain. The study will assess the safety of administering multiple doses of XARTEMIS XR in this population.

ELIGIBILITY:
Inclusion criteria:

1. Male or nonpregnant, nonlactating females between 12 and 17 years of age.
2. Minimum weight of 100 pounds (45 kg); body mass index (BMI) >5% and <95% for their age.
3. Moderate or severe acute pain [as determined from the Numerical Pain Rating scale (NPRS)]; must have a level of 4 or more) after surgical procedure requiring hospitalization.
4. If, of child-bearing/reproductive potential, must abstain from unprotected sexual activity during study and 2 weeks after study exit.
5. Females of childbearing potential must have negative pregnancy test.
6. Subject's legally authorized representative (eg, parent, legal guardian) must sign a parental permission/informed consent and subject must sign an assent.
7. Subject and subject's parent/legal guardian must be able to read, understand, and follow study procedures and requirements and communicate meaningfully in English.

Exclusion criteria:

1. Subject is from a vulnerable population (including mentally disabled children), other than a pediatric population.
2. Subject requires surgery that could influence the study outcome.
3. Abnormal electrocardiogram (ECG).
4. Screening pulse oximetry reading of <95% while awake.
5. Has presence of human immunodeficiency virus (HIV) or indications of hepatitis A, B or C.
6. Lab values greater than 2 times the upper limit of normal.
7. History of renal disease or bleeding or clotting disorders or conditions.
8. Known or suspected alcoholism, marijuana or illicit drug abuse or misuse within 2 years before screening.
9. Smoked or used nicotine-containing products within 6 months prior to screening.
10. Psychiatric disorders, such as major depression disorder, anxiety disorders, or psychotic disorders within 6 months prior to screening. A history of attention deficit hyperactivity disorder requiring medication is acceptable.
11. Diagnosis of epilepsy or other seizure disorder.
12. Previous cardiothoracic surgery.
13. Conditions which might be specifically contraindicated or require caution while using OC, APAP, and/or ibuprofen.
14. Drug allergy, hypersensitivity, or intolerance including OC, APAP, ibuprofen or excipients, or any opioid drug product.
15. Donated or had significant loss of whole blood (480 mL or more) within 30 days of or plans to donate blood or plasma during the course of the study.
16. Pathologic, iatrogenic or surgical condition that would compromise subject's ability to swallow, absorb, metabolize, or excrete XARTEMIS XR.
17. History of a GI event within 6 months prior to screening.
18. Subject has used any product containing OC or APAP within 48 hours prior to the first dose of XARTEMIS XR.
19. Any other medical condition, abnormal vital sign (blood pressure, pulse rate, respiratory rate), body temperature, pulse oximetry; or any physical examination or ECG finding at screening which would preclude safe participation in a clinical study.
20. Received any investigational product or device within 30 days before screening, or is scheduled to receive an investigational device or another investigational drug during the course of this study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2017-04-26 (Actual); Study Completion 2017-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Mallinckrodt
Locations (2):
- United States (2):
  - Duke University Health Systems, Durham, North Carolina
  - University of Pittsburgh Medical Center, University of Pittsburgh Physicians, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from November 20, 2015 to April 26, 2017 and enrolled participants from the United States.
Groups:
- XARTEMIS XR: XARTEMIS XR is a combination of oxycodone and acetaminophen administered to postsurgical adolescent participants with moderate to severe acute pain.
Period: Overall Study
Arm/Group | XARTEMIS XR
Started | 23
Completed | 0
Not Completed | 23
Not completed — Withdrawal by Subject | 1
Not completed — Withdrawal by Caregiver | 8
Not completed — Pain Score <4 | 1
Not completed — Emesis | 3
Not completed — Adverse Event | 3
Not completed — Protocol Violation | 1
Not completed — Physician Decision | 1
Not completed — Trial terminated by sponsor | 5

BASELINE CHARACTERISTICS:
Population: The Safety population included all participants who enrolled in the study and received any quantity of XARTEMIS XR.
Arm/Group | XARTEMIS XR
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.7 (1.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Reach Steady State
Description: The time to reach steady state in participants who received all 5 doses
Time Frame: within 60 hours
Population: Steady-state pharmacokinetic (PK) parameters were to be determined for those participants administered all 5 doses. However, no participant received all 5 doses; therefore, steady state PK parameters were not derived.
Groups:
- XARTEMIS XR: All participants received XARTEMIS XR
  XARTEMIS XR: XARTEMIS XR (7.5 mg oxycodone hydrochloride and 325 mg acetaminophen) Extended-Release Tablets
Arm/Group | XARTEMIS XR
Number analyzed (Participants) | 0

2. Primary Outcome: Area Under the Concentration-time Curve (AUC) From Time Zero (AUC0) to the Time of the Last Quantifiable Plasma Sample (AUClast)
Description: Elimination constant estimates required for the calculation of the planned AUC0-12 hours were not available. AUClast therefore provided the best available measure of exposure, effectively representing AUC0-12 hours for both moieties. While considered the best available measure, it also remains inaccurate because of the extended-release formulation and the lack of data beyond the 12.08-hour time point.
Time Frame: within approximately 12 hours (12.08 hours)
Population: PK population
Measure: Median (Full Range); unit: ng*hr/mL
Groups:
- Oxycodone: Pharmacokinetics of oxycodone were collected for 12 hours after dosing of XARTEMIS XR on Study Day 1
- Acetaminophen: Pharmacokinetics of acetaminophen were collected for 12 hours after dosing of XARTEMIS XR on Study Day 1
Arm/Group | Oxycodone | Acetaminophen
Number analyzed (Participants) | 18 | 18
ng*hr/mL | 76.8 [25.85 to 173.59] | 20571.4 [10195.17 to 33714.50]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: The highest concentration of study drug within 12 hours.
Time Frame: within approximately 12 hours (12.08 hours)
Population: PK population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oxycodone | Acetaminophen
Number analyzed (Participants) | 18 | 18
ng/mL | 12.8 (4.6) | 2886.1 (881.68)

4. Primary Outcome: Apparent Plasma Terminal Drug Elimination Half-life (T1/2)
Description: PK parameters are determined after a single administration of study drug on Day 1. Plasma concentrations that are below the level of quantification (BLQ) are set to 0 before Tmax, with the exception that a BLQ value occurring between measurable concentrations is set to missing. BLQ values that occur after Tmax are set to missing.
Time Frame: within approximately 12 hours (12.08 hours)
Population: PK population with BLQ values set to missing
Measure: Median (Full Range); unit: hours
Arm/Group | Oxycodone | Acetaminophen
Number analyzed (Participants) | 10 | 16
hours | 0.52 [0.00 to 2.83] | 0.00 [0.00 to 0.97]

5. Primary Outcome: Time of Maximum Observed Plasma Concentration (Tmax)
Description: The time at which the maximum plasma concentration (Cmax) is reached.
Time Frame: within approximately 12 hours (12.08 hours)
Population: PK population.
Measure: Median (Full Range); unit: hour
Arm/Group | Oxycodone | Acetaminophen
Number analyzed (Participants) | 18 | 18
hour | 7.9 [3.92 to 12.08] | 4.03 [2.07 to 12.08]

ADVERSE EVENTS:
Time Frame: Up to 17 months.
Description: A treatment-emergent adverse event (TEAE) is defined as an evat that emerges during treatment having been absent pre-treatment or worsens relative to the pre-treatment state. Any TEAE determined as possibly related or related to the study drug is considered a treatment-related TEAE. All serious adverse events are reported, as well as all treatment-related TEAEs.
Arm/Group | XARTEMIS XR
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 3/23
Other Adverse Events (participants affected / at risk) | 7/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XARTEMIS XR (N=23)
Severe pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Moderate Constipation (Gastrointestinal disorders) | 1
Severe delirium (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XARTEMIS XR (N=23)
Constipation (Gastrointestinal disorders) | 3
Pruritis (Skin and subcutaneous tissue disorders) | 2
Asthenia (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators will be part of the primary publication. Each investigator may publish on the data from subjects enrolled at their site after the initial publication has been submitted.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT02508935/Prot_SAP_000.pdf